CLINICAL TRIAL: NCT03930797
Title: Addressing Sexual Concerns in Breast Cancer Survivors: Randomized Controlled Trial of a Novel Couple-Based Intervention
Brief Title: Coping Together After Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 18-1025; 1R01CA222124-01A1 (NIH)
Record Dates: First submitted 2019-04-24; First posted 2019-04-29 (Actual); Results first posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intimacy Enhancement (Experimental): Participants attend four sessions (60-75 minutes) consisting of education and skills training to enhance physical and emotional intimacy.
  Interventions: Behavioral: Intimacy Enhancement
- Living Healthy Together (Active Comparator): Participants attend four sessions (60-75 minutes) consisting of information and support across a range of breast cancer-related topics.
  Interventions: Behavioral: Living Healthy Together

INTERVENTIONS:
Behavioral: Intimacy Enhancement — The IE intervention is grounded in cognitive behavioral couple therapy and sex therapy, and includes education and skills training with a focus on the following major topics: understanding effects of breast cancer on sex and intimacy; goal-setting; communication skills; problem-solving and engaging in activities to build intimacy; identifying and restructuring negative or inflexible thoughts; and planning ahead and preparing for challenges. Participants will be asked to participate in written and behavioral activities at home between sessions to strengthen skills acquisition.
  Arms: Intimacy Enhancement
Behavioral: Living Healthy Together — The Living Healthy Together (LHT) intervention focuses on delivering education and support to breast cancer survivors and their partners across a range of topics including social support, sleep and fatigue, stress and stress management, nutrition, and physical activity. Participants will be asked to engage actively with the material and to review readings and intervention material between sessions.
  Arms: Living Healthy Together

SUMMARY:
The objective of the proposed study is to evaluate an Intimacy Enhancement (IE) intervention in 120 female early stage breast cancer survivors reporting sexual concerns and their intimate partners (240 total participants). Couples will be randomized 1:1 to receive either the IE intervention or to an information and support condition (Living Healthy Together). The investigators will evaluate intervention effects on patient and partner sexual, relationship, and psychological outcomes.

DETAILED DESCRIPTION:
Over half of breast cancer survivors experience sexual concerns resulting from physical changes due to breast surgery, chemotherapy, and hormonal therapies; emotional changes; and relationship difficulties. In contrast with many aspects of quality of life (QOL) that tend to improve over time for breast cancer survivors, sexual concerns often persist for years. As a result, many breast cancer survivors and their partners may wish to resume a satisfying intimate relationship after treatment ends but encounter difficulties in doing so. Sexual concerns often go unaddressed, can lead to clinically significant psychological distress, and have a negative impact on survivors' relationships and quality of life. Thus, addressing sexual concerns and improving sexual function is of critical importance to the long-term adjustment of these survivors. Given the central role of the intimate relationship in breast cancer survivors' sexual experiences, a couple-based intervention that systematically involves the partner may be a highly effective approach for addressing these concerns and improving function. Yet randomized controlled trials evaluating the efficacy of a couple-based intervention targeting sexual function for breast cancer survivors are lacking. In this study, the investigators plan to evaluate a four-session telephone couple-based intervention that provides education and training in cognitive and behavioral skills to help couples cope with sexual concerns and enhance their intimate relationship, called Intimacy Enhancement (IE).

The specific aims of this study are (1) to evaluate whether the IE intervention will lead to a significantly greater increase in patient sexual function from pre-treatment to post-treatment and 3- and 6-month follow-ups compared to the LHT condition; (2) to evaluate whether the IE intervention will lead to significantly greater improvements in partner sexual function, patient sexual distress, patient/partner relationship intimacy/quality, and psychological distress from pre-treatment to post-treatment and at 3- and 6-month follow-ups, compared to the LHT condition; (3) to evaluate whether increases from pre- to post-treatment in patient sexual communication and self-efficacy for coping with sexual concerns mediate the beneficial effects of the IE intervention on patient sexual function at 3- and 6-month follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* Patient is female
* Patient age 18 years or older
* Patient has a medically confirmed diagnosis of non-recurrent breast cancer (Stages T1-T4, N0-N1, M0)
* Patient completed active treatment (e.g., chemotherapy, radiation therapy, surgery, immunotherapy) 6 months-5 years ago (current use of endocrine therapy is acceptable)
* Patient is currently in a partnered relationship that could involve sexual activity
* Partner or spouse is 18 years or older
* Patient lives with a romantic partner for at least 6 months
* Patient has a score of at least 3 on Patient Care Monitor Sexual Concerns screening item

Exclusion Criteria:

* Patient or partner is not able to speak and read English, as stated in medical record, as observed by study team member or in self-report
* Patient or partner ECOG Performance score > 2 OR medically unable to participate as judged by physician/in medical record or by self-report
* Patient or partner has a hearing impairment
* Patient and partner do not have reliable telephone access
* Patient has overt cognitive dysfunction or psychiatric disturbance such as suicidal ideation or severe mental illness, as observed or judged by the researcher, physician or referring source, or self-report
* Patient past or current history of any cancer other than non-melanoma skin cancer, including prior breast cancer
* Patient is currently participating in couple/marital therapy
* Patient is currently pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2019-05-24 (Actual); Primary Completion 2023-04-14 (Actual); Study Completion 2023-04-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reese JB, Zimmaro LA, Lepore SJ, Sorice KA, Handorf E, Daly MB, Schover LR, Kashy D, Westbrook K, Porter LS. Evaluating a couple-based intervention addressing sexual concerns for breast cancer survivors: study protocol for a randomized controlled trial. Trials. 2020 Feb 12;21(1):173. doi: 10.1186/s13063-019-3975-2. PMID 32051002

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants receive one telephone intervention or the other (IE or LHT); due to this, randomization occurs after the first telephone session is already scheduled so as not to waste randomization slots on couples who have no intention of following through with sessions.
  As such, participants may be "lost" prior to randomization if they complete consent/baseline but never schedule their first telephone session.
Period: Overall Study
Arm/Group | Intimacy Enhancement | Living Healthy Together
Started | 122 | 118
Completed | 119 | 108
Not Completed | 3 | 10
Not completed — Lost to Follow-up | 3 | 10

BASELINE CHARACTERISTICS:
Population: We present data separately for patients and partners, even though dyads were assigned to the same study arm, as our outcomes are patient- and partner-specific.
Groups:
- Patient Intimacy Enhancement; Partner Intimacy Enhancement: Participants attend four sessions (60-75 minutes) consisting of education and skills training to enhance physical and emotional intimacy.
  Intimacy Enhancement: The IE intervention is grounded in cognitive behavioral couple therapy and sex therapy, and includes education and skills training with a focus on the following major topics: understanding effects of breast cancer on sex and intimacy; goal-setting; communication skills; problem-solving and engaging in activities to build intimacy; identifying and restructuring negative or inflexible thoughts; and planning ahead and preparing for challenges. Participants will be asked to participate in written and behavioral activities at home between sessions to strengthen skills acquisition.
- Patient Living Healthy Together; Partner Living Healthy Together: Participants attend four sessions (60-75 minutes) consisting of information and support across a range of breast cancer-related topics.
  Living Healthy Together: The Living Healthy Together (LHT) intervention focuses on delivering education and support to breast cancer survivors and their partners across a range of topics including social support, sleep and fatigue, stress and stress management, nutrition, and physical activity. Participants will be asked to engage actively with the material and to review readings and intervention material between sessions.
- Total: Total of all reporting groups
Arm/Group | Patient Intimacy Enhancement | Patient Living Healthy Together | Partner Intimacy Enhancement | Partner Living Healthy Together | Total
Number analyzed (Participants) | 61 | 59 | 61 | 59 | 240
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.39 (9.60) | 51.12 (9.97) | 52.26 (10.37) | 52.64 (11.15) | 51.60 (10.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 59 | 0 | 3 | 123
  Male | 0 | 0 | 61 | 56 | 117
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 1 | 3
  Not Hispanic or Latino | 60 | 57 | 60 | 58 | 235
  Unknown or Not Reported | 0 | 2 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 1 | 1 | 0 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 8 | 7 | 8 | 8 | 31
  White | 52 | 48 | 53 | 48 | 201
  More than one race | 0 | 2 | 0 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 61 | 59 | 61 | 59 | 240
Level of Sexual Concerns [Mean (Standard Deviation); unit: units on a scale] — Level of sexual concerns for patients on a scale of 0-10, with 0 indicating no sexual concerns and 10 indicating severe sexual concerns. Measure administered to patients only. Population: Measure given to patient participants only.
  units on a scale
    number analyzed (Participants) | 61 | 59 | 0 | 0 | 120
    (all) | 6.18 (1.90) | 6.32 (1.99) |  |  | 6.25 (1.94)
Length of Relationship (years) [Mean (Standard Deviation); unit: years] — Population: Measure given to patient participants only
  years
    number analyzed (Participants) | 61 | 59 | 0 | 0 | 120
    (all) | 21.65 (11.66) | 20.54 (12.29) |  |  | 21.10 (11.94)
Time Since Diagnosis (months) [Mean (Standard Deviation); unit: months] — Population: Measure given to patient participants only
  months
    number analyzed (Participants) | 61 | 59 | 0 | 0 | 120
    (all) | 28.69 (14.77) | 31.32 (13.02) |  |  | 29.98 (13.94)
Time Since Treatment Completion (months) [Mean (Standard Deviation); unit: months] — Population: Measure given to patient participants only
  months
    number analyzed (Participants) | 61 | 59 | 0 | 0 | 120
    (all) | 20.40 (13.04) | 23.55 (12.52) |  |  | 21.95 (12.83)
Education [Count of Participants; unit: Participants]
  Less than high school | 0 | 0 | 1 | 1 | 2
  High school | 6 | 8 | 13 | 11 | 38
  Some college | 19 | 12 | 14 | 13 | 58
  College degree | 23 | 18 | 16 | 21 | 78
  Graduate school | 13 | 21 | 17 | 13 | 64
Employment [Count of Participants; unit: Participants]
  Employed full time/part time | 42 | 43 | 48 | 45 | 178
  Unemployed/on disability | 15 | 12 | 5 | 5 | 37
  Retired | 4 | 4 | 8 | 9 | 25
Relationship Status [Count of Participants; unit: Participants] — Population: Measure given to patient participants only. One IE patient and one LHT patient did not respond to this item on the survey.
  Participants
    number analyzed (Participants) | 60 | 58 | 0 | 0 | 118
    Married | 58 | 49 |  |  | 107
    Cohabitating, not married | 2 | 9 |  |  | 11
Sexual Orientation [Count of Participants; unit: Participants]
  Heterosexual/straight | 59 | 56 | 61 | 55 | 231
  Homosexual/lesbian/gay | 0 | 2 | 0 | 1 | 3
  Bisexual | 2 | 1 | 0 | 3 | 6
Patient Clinical Tumor Stage [Count of Participants; unit: Participants] — Clinical tumor stage reflects the estimated tumor size and/or amount of spread into nearby structures at diagnosis. Higher tumor stage (e.g., cT4) indicates a larger tumor or spread and is associated with worse outcomes. Population: Data available for patient participants only
  Participants
    number analyzed (Participants) | 61 | 59 | 0 | 0 | 120
    cT1 | 39 | 36 |  |  | 75
    cT2 | 16 | 15 |  |  | 31
    cT3 | 4 | 6 |  |  | 10
    cT4 | 2 | 2 |  |  | 4
Patient Surgery Received [Count of Participants; unit: Participants] — Population: Data available for patient participants only
  Participants
    number analyzed (Participants) | 61 | 59 | 0 | 0 | 120
    Lumpectomy | 24 | 25 |  |  | 49
    Mastectomy with reconstruction | 24 | 22 |  |  | 46
    Mastectomy without reconstruction | 13 | 12 |  |  | 25
Patient Radiotherapy Received [Count of Participants; unit: Participants] — Population: Data available for patient participants only
  Participants
    number analyzed (Participants) | 61 | 59 | 0 | 0 | 120
    Radiotherapy received | 48 | 45 |  |  | 93
    Radiotherapy not received | 13 | 14 |  |  | 27
Patient Chemotherapy Received [Count of Participants; unit: Participants] — Population: Data available for patient participants only
  Participants
    number analyzed (Participants) | 61 | 59 | 0 | 0 | 120
    Chemotherapy received | 40 | 31 |  |  | 71
    Chemotherapy not received | 21 | 28 |  |  | 49
Patient Immunotherapy Received [Count of Participants; unit: Participants] — Population: Data available for patient participants only
  Participants
    number analyzed (Participants) | 61 | 59 | 0 | 0 | 120
    Immunotherapy received | 13 | 12 |  |  | 25
    Immunotherapy not received | 48 | 47 |  |  | 95
Patient Endocrine Therapy Received [Count of Participants; unit: Participants] — Population: Data available for patient participants only
  Participants
    number analyzed (Participants) | 61 | 59 | 0 | 0 | 120
    Endocrine therapy received | 44 | 48 |  |  | 92
    Endocrine therapy not received | 17 | 11 |  |  | 28
Patient Ovarian Suppression therapy Received [Count of Participants; unit: Participants] — Population: Data available for patient participants only
  Participants
    number analyzed (Participants) | 61 | 59 | 0 | 0 | 120
    Ovarian suppression received | 14 | 11 |  |  | 25
    Ovarian suppression not received | 47 | 48 |  |  | 95
Patient Currently Receiving Endocrine/Ovarian Suppression Therapy [Count of Participants; unit: Participants] — Population: Data available for patient participants only
  Participants
    number analyzed (Participants) | 61 | 59 | 0 | 0 | 120
    Currently receiving endocrine/ovarian suppression therapy | 45 | 43 |  |  | 88
    Not currently receiving endocrine/ovarian suppression therapy | 16 | 16 |  |  | 32
Patient Gynecologic Surgeries [Count of Participants; unit: Participants] — Population: Data available for patient participants only
  Participants
    number analyzed (Participants) | 61 | 59 | 0 | 0 | 120
    Oophorectomy | 18 | 11 |  |  | 29
    Hysterectomy | 15 | 9 |  |  | 24
    No gynecologic surgery | 28 | 39 |  |  | 67
Patient Menopausal Status [Count of Participants; unit: Participants] — Population: Data available for patient participants only
  Participants
    number analyzed (Participants) | 61 | 59 | 0 | 0 | 120
    Post-menopausal | 46 | 34 |  |  | 80
    Pre-menopausal | 13 | 16 |  |  | 29
    Peri-menopausal | 2 | 9 |  |  | 11

OUTCOME MEASURES:

1. Primary Outcome: Change in Self-Reported Patient Sexual Function
Description: Patients' self-reported sexual function will be measured using the 19-item Female Sexual Function Index (FSFI).Total scale scores range from 2 to 36, with higher scores indicating higher functioning. Mean change scores will be reported: positive mean change scores indicate increase in sexual functioning over time while negative mean change scores indicate decrease in sexual functioning over time.
Time Frame: Baseline up to 6 weeks
Population: Only patient participants' data was analyzed for this aim. Of 61 IE patients, one did not return the 6-week follow-up assessment. Of 59 LHT patients, 4 did not return the 6-week follow-up assessment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intimacy Enhancement | Living Healthy Together
Number analyzed (Participants) | 60 | 55
score on a scale | 6.41 (7.35) | 0.90 (6.99)

2. Secondary Outcome: Change in Self-Reported Partner Sexual Function
Description: Partners' (male) self-reported sexual function will be measured using the 15-item International Index of Erectile Function (IIEF). Total scale scores range from 1 to 75, with higher scores indicating a higher level of sexual functioning. Change in mean male partner IIEF score over time will be reported. Positive mean change scores indicate increase in sexual functioning.
Time Frame: Baseline up to 6 weeks
Population: Only male partner participants' data were included in this analysis. Of 61 IE partners, one did not complete the 6-week follow-up assessment. Of 59 LHT partners, 2 were female, 3 did not return the 6-week follow-up assessment, and 1 did not have sufficient data to calculate a change score.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intimacy Enhancement | Living Healthy Together
Number analyzed (Participants) | 60 | 53
score on a scale | 2.48 (12.92) | 1.00 (12.19)

3. Secondary Outcome: Change in Self-Reported Patient Sexual Distress
Description: Patient sexual distress will be measured using the 13-item Female Sexual Distress Scale-Revised (FSDS-R). Total scale scores range from 0 to 52. Higher scores indicate higher levels of sexual distress. Change in patient mean sexual distress score over time will be reported. Negative mean change scores indicate decrease in sexual distress.
Time Frame: Baseline up to 6 weeks
Population: Only patient participants' data were used for this analysis. Of 61 IE patients, one did not complete the 6-week follow-up assessment. Of 59 LHT patients, 4 did not complete the 6-week follow-up assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intimacy Enhancement | Living Healthy Together
Number analyzed (Participants) | 60 | 55
score on a scale | -7.82 (9.49) | -4.40 (8.98)

4. Secondary Outcome: Change in Patients' Self-Reported Relationship Intimacy
Description: Patient self-reported relationship intimacy will be measured using the 17-item Miller Social Intimacy Scale (MSIS). This scale assesses emotional intimacy, closeness and trust toward an individual's partner. Scores range from 17 to 170, with higher scores indicating higher levels of intimacy. Change in patient mean relationship intimacy score over time will be reported. Positive mean change scores indicate increase in relationship intimacy.
Time Frame: Baseline up to 6 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intimacy Enhancement | Living Healthy Together
Number analyzed (Participants) | 60 | 55
score on a scale | 7.58 (15.96) | 5.85 (12.63)

5. Secondary Outcome: Change in Partners' Self-Reported Relationship Intimacy
Description: Partner self-reported relationship intimacy will be measured using the 17-item Miller Social Intimacy Scale (MSIS). This scale assesses emotional intimacy, closeness and trust toward an individual's partner. Scores range from 17 to 170, with higher scores indicating higher levels of intimacy. Change in patient mean relationship intimacy score over time will be reported. Positive mean change scores indicate increase in relationship intimacy.
Time Frame: Baseline up to 6 weeks
Population: Only partner participants' data were used for this analysis. Of 61 IE partners, one did not complete the 6-week follow-up assessment. Of 59 LHT partners, 4 did not complete the 6-week follow-up assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intimacy Enhancement | Living Healthy Together
Number analyzed (Participants) | 60 | 55
score on a scale | 6.35 (13.80) | 5.77 (14.37)

6. Secondary Outcome: Change in Patients' Self-Reported Relationship Quality
Description: Patient self-reported relationship quality will be measured using the 7-item Dyadic Adjustment Scale (DAS-7). Total scale scores range from 0 to 36. Higher scores indicate higher relationship quality. Change in mean relationship quality score over time will be reported. Positive mean change scores indicate increase in relationship quality.
Time Frame: Baseline up to 6 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intimacy Enhancement | Living Healthy Together
Number analyzed (Participants) | 60 | 55
score on a scale | 1.20 (4.34) | 2.49 (4.59)

7. Secondary Outcome: Change in Partners' Self-Reported Relationship Quality
Description: Partner self-reported relationship quality will be measured using the 7-item Dyadic Adjustment Scale (DAS-7). Total scale scores range from 0 to 36. Higher scores indicate higher relationship quality. Change in mean relationship quality score over time will be reported. Positive mean change scores indicate increase in relationship quality.
Time Frame: Baseline up to 6 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intimacy Enhancement | Living Healthy Together
Number analyzed (Participants) | 60 | 55
score on a scale | 1.65 (4.26) | 1.27 (3.69)

8. Secondary Outcome: Change in Patients' Self-Reported Anxiety
Description: Patients' self-reported anxiety will be measured using the 7-item Generalized Anxiety Disorder scale (GAD-7). Total scale scores range from 0 to 21. Higher scores indicate higher levels of anxiety. Change in mean anxiety score over time will be reported. Negative mean change scores indicate decrease in anxiety.
Time Frame: Baseline up to 6 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intimacy Enhancement | Living Healthy Together
Number analyzed (Participants) | 60 | 55
score on a scale | -0.70 (3.25) | 0.07 (3.83)

9. Secondary Outcome: Change in Partners' Self-Reported Anxiety
Description: Partners' self-reported anxiety will be measured using the 7-item Generalized Anxiety Disorder scale (GAD-7). Total scale scores range from 0 to 21. Higher scores indicate higher levels of anxiety. Change in mean anxiety score over time will be reported. Negative mean change scores indicate decrease in anxiety.
Time Frame: Baseline up to 6 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intimacy Enhancement | Living Healthy Together
Number analyzed (Participants) | 60 | 55
score on a scale | -0.98 (2.95) | 0.27 (2.80)

10. Secondary Outcome: Change in Patients' Self-Reported Depressive Symptoms
Description: Patients' self-reported depression will be measured using the 9-item Patient Health Questionnaire (PHQ-9). Total scale scores range from 0 to 27. Higher scores indicate higher levels of depression. Change in mean depression score over time will be reported. Negative mean change scores indicate decrease in depression.
Time Frame: Baseline up to 6 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intimacy Enhancement | Living Healthy Together
Number analyzed (Participants) | 60 | 55
score on a scale | -0.99 (4.36) | -0.74 (3.31)

11. Secondary Outcome: Change in Partners' Self-Reported Depressive Symptoms
Description: Partners' self-reported depression will be measured using the 9-item Patient Health Questionnaire (PHQ-9). Total scale scores range from 0 to 27. Higher scores indicate higher levels of depression. Change in mean depression score over time will be reported. Negative mean change scores indicate decrease in depression.
Time Frame: Baseline up to 6 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intimacy Enhancement | Living Healthy Together
Number analyzed (Participants) | 60 | 55
score on a scale | -0.61 (2.47) | -0.16 (4.10)

ADVERSE EVENTS:
Time Frame: Adverse events were tracked over the course of study participation (6 months).
Groups:
- Intimacy Enhancement Patients; Intimacy Enhancement Partners: Participants attend four sessions (60-75 minutes) consisting of education and skills training to enhance physical and emotional intimacy.
  Intimacy Enhancement: The IE intervention is grounded in cognitive behavioral couple therapy and sex therapy, and includes education and skills training with a focus on the following major topics: understanding effects of breast cancer on sex and intimacy; goal-setting; communication skills; problem-solving and engaging in activities to build intimacy; identifying and restructuring negative or inflexible thoughts; and planning ahead and preparing for challenges. Participants will be asked to participate in written and behavioral activities at home between sessions to strengthen skills acquisition.
- Living Healthy Together Patients; Living Healthy Together Partners: Participants attend four sessions (60-75 minutes) consisting of information and support across a range of breast cancer-related topics.
  Living Healthy Together: The Living Healthy Together (LHT) intervention focuses on delivering education and support to breast cancer survivors and their partners across a range of topics including social support, sleep and fatigue, stress and stress management, nutrition, and physical activity. Participants will be asked to engage actively with the material and to review readings and intervention material between sessions.
Arm/Group | Intimacy Enhancement Patients | Living Healthy Together Patients | Intimacy Enhancement Partners | Living Healthy Together Partners
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/59 | 0/61 | 0/59
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/59 | 0/61 | 0/59
Other Adverse Events (participants affected / at risk) | 3/61 | 6/59 | 2/61 | 4/59
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intimacy Enhancement Patients (N=61) | Living Healthy Together Patients (N=59) | Intimacy Enhancement Partners (N=61) | Living Healthy Together Partners (N=59)
Self-reported distress (Psychiatric disorders) | 3 | 6 | 2 | 4 — Any report of thoughts of self harm/being better off dead on the Patient Health Questionnaire, given at all time points.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-14): https://cdn.clinicaltrials.gov/large-docs/97/NCT03930797/Prot_SAP_000.pdf